CLINICAL TRIAL: NCT00147719
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study of the Efficacy and Safety of WelChol® in Type 2 Diabetics With Inadequate Glycemic Control on Metformin Monotherapy or Metformin Therapy in Combination With Other Oral Anti-Diabetic Agents
Brief Title: WelChol® With Metformin in Treating Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WEL-301
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Colesevelam Hydrochloride

INTERVENTIONS:
Drug: Colesevelam hydrochloride

SUMMARY:
The purpose of the study is to see how safe and effective and tolerable the use of colesevelam hydrochloride is for type 2 diabetes when added to metformin alone or in combination with other anti-diabetic drugs.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years, inclusive
* Diagnosed with type 2 diabetes
* Hemoglobin (HbA1c) between 7.5% to 9.5%
* Prescribed an ADA accepted diet
* Receiving stable dose of metformin alone or in combination with other oral anti-diabetic medications for 90 days before Visit 1

Exclusion Criteria:

* History of type 1 diabetes or ketoacidosis
* History of chronic (more than 2 months) insulin therapy or the initiation of insulin for chronic treatment
* History of pancreatitis
* Uncontrolled hypertension
* Recent severe cardiovascular disease
* Allergy or toxic response to colesevelam or any of its components
* Body mass index (BMI) >45 kg/m2

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2004-06; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
To assess the additional lowering of HbA1C achieved by addition of colesevelam hydrochloride to current antidiabetic therapy

SECONDARY OUTCOMES:
To assess the fasting plasma glucose and fructosamine lowering effect;
To assess the glycemic control response rate;
To assess the improvement in insulin sensitivity;
To assess the effect on high sensitivity C-reactive protein;
To assess the improvement in lipids, and lipoproteins;
To assess the safety and tolerability of colesevelam hydrochloride when added on to current therapy

CONTACTS AND LOCATIONS:
Locations (48):
- United States (46):
  - CRO, Jonesboro, Arkansas
  - Beverly Hills, California
  - Carmichael, California
  - Fresno, California
  - Irvine, California
  - La Jolla, California
  - Los Gatos, California
  - San Diego, California
  - Spring Valley, California
  - West Hills, California
  - Washington D.C., District of Columbia
  - Coco Beach, Florida
  - Largo, Florida
  - Miami, Florida
  - Pembroke Pines, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Evansville, Indiana
  - Louisville, Kentucky
  - Detroit, Michigan
  - Troy, Michigan
  - Edina, Minnesota
  - Chesterfield, Missouri
  - Bozeman, Montana
  - Butte, Montana
  - Las Vegas, Nevada
  - Rochester, New York
  - Charlotte, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Lyndhurst, Ohio
  - Marion, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Beaver, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Morristown, Tennessee
  - Corpus Christi, Texas
  - Dallas, Texas
  - Pharr, Texas
  - San Antonio, Texas
  - Arlington, Virginia
  - Richmond, Virginia
- Mexico City, Mexico
- Lima, Peru

REFERENCES:
- [Derived] Bays HE, Goldberg RB, Truitt KE, Jones MR. Colesevelam hydrochloride therapy in patients with type 2 diabetes mellitus treated with metformin: glucose and lipid effects. Arch Intern Med. 2008 Oct 13;168(18):1975-83. doi: 10.1001/archinte.168.18.1975. PMID 18852398